CLINICAL TRIAL: NCT01116388
Title: A Study to Assess the Role of a Gluten Free-Casein Free Diet in the Dietary Management of Autism Associated Gastrointestinal Disorders
Brief Title: A Study to Assess the Role of a Gluten Free-dairy Free (GFCF) Diet in the Dietary Management of Autism Associated Gastrointestinal Disorders
Acronym: GFCF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Nutricia North America (Industry)
Responsible Party: Principal Investigator, Harland S. Winter, MD, Director, Pediatric Inflammatory Bowel Disease Center, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008-P-002385
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Autism; Gastrointestinal Symptoms
Keywords: Autism; Gastrointestinal Disorders; Food Allergy; Gluten free, casein free diet; Diarrhea; Constipation; Reflux; Abdominal pain; Pain after eating; Self injurious behavior
MeSH Terms: conditions — Autistic Disorder; Gastrointestinal Diseases; Food Hypersensitivity; Diarrhea; Constipation; Gastroesophageal Reflux; Abdominal Pain; Self-Injurious Behavior | interventions — Caseins; Milk Proteins; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- test product (Other): product free of gluten and casein
  Interventions: Other: GFCF product with GFCF diet
- control product (Other): product containing gluten and milk protein
  Interventions: Other: product containing gluten and casein (milk protein) with GFCF diet

INTERVENTIONS:
Other: GFCF product with GFCF diet — Group I: will receive the test product (product free of gluten and casein) with GFCF Diet for the 1st 6-weeks.
  Group II: will receive the test product (product free of gluten and casein) with GFCF diet for the 2nd 6-weeks.
  Other Names: test product; GFCF; gluten free- casein free diet
  Arms: test product
Other: product containing gluten and casein (milk protein) with GFCF diet — Group I: will receive the control product (product containing gluten and casein) with the GFCF diet for the 2nd 6-weeks.
  Group II: will receive the control product (product containing gluten and casein) with the GFCF diet for the 1st 6-weeks
  Other Names: control product; product containing gluten and casein; GFCF diet
  Arms: control product

SUMMARY:
Doctors at MassGeneral Hospital for Children (MGHfC) are doing a research study to learn if a gluten free-dairy free (GFCF) diet is helpful in improving gastrointestinal symptoms associated with autism.

Hypothesis: The gluten free/casein free diet (GFCF) will result in a higher proportion of subjects having reduction in gastrointestinal (GI) symptoms associated with autism spectrum disorders (ASD).

Primary Study Objective:

* To assess the effect of a GFCF diet on GI symptoms associated with ASD.

Secondary Objectives:

* To assess if improvements in GI symptoms result in improvements in autistic behavior when using a GFCF diet in the dietary management of GI symptoms associated with ASD
* To determine the nutritional impact of a GFCF restrictive diet
* To assess the role of food allergies in the manifestation of GI symptoms

This is a 14-week study that requires between 5 & 9 office visits. All study related activities -including physical exams, blood samples and allergy testing - and an amino acid based supplement drink, are at no cost. Research study visits will take place at MGHfC in Boston, or at Newton Wellesley Hospital in Newton, or at Lurie Center/LADDERS in Lexington.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent / Assent, as applicable must be signed prior to executing any study related procedure
* Children, male or female, 2 to 17 years old (inclusive)
* Confirmed diagnosis of ASD according to the diagnostic measures:

  * DSM-IV Symptom Checklist
  * Autism Diagnostic Observation Schedule(ADOS)&/or Autism Diagnostic Interview Revised(ADI-R)within 18 months prior to entry into the study
* Subjects must present with a current history of at least two of the following persistent GI symptoms as confirmed by the study physician:

  * Diarrhea, as characterised by three or more loose stools a day for at least 8 out of 14 days
  * Constipation as characterised by less than 3 bowel movements per week, for at least a 2-week period
  * Esophageal reflux, as characterised by 3 or more episodes of regurgitation per day on 10 out of 14 days
  * Abdominal pain manifested as pain after eating or self injurious behavior on at least 8 out of 14 days
  * Suspected food allergy which is confirmed by a physician, as characterized as a recurrent reaction or association with specific foods
* Subject able to consume 3 tablespoons of study powder mixed in food daily for 12 weeks

Exclusion Criteria:

* Children with a history of anaphylaxis to dietary milk and wheat proteins
* Children with severe concurrent illness
* Children who are prescribed systemic steroids
* Children currently receiving chelation therapy, hyperbaric or antifungal treatment within 1 month of entry into the study and during the study period.
* Children with a confirmed diagnosis of celiac disease
* Subjects who have previously tried dietary elimination of casein and gluten for at least 1 month period and failed to demonstrate a response by parent perception
* Children who are unable to consume 3 tablespoons of study powder mixed in food daily for 12 weeks daily

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2010-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
A study to assess the role of a gluten free-casein free diet in the dietary management of autism associated gastrointestinal disorders | 12 weeks
  The effect of a GFCF diet on the dietary management of GI symptoms associated with autism is the primary outcome measure in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Harland S Winter, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Baylor College of Medicine / Texas Children's Hospital, Houston, Texas